CLINICAL TRIAL: NCT00781729
Title: Phase 2 Study of Yoga for Excess Thoracic Curvature.
Brief Title: Yoga for Kyphosis Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Gail A. Greendale, MD, Geffen SOM at UCLA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AG030448-01A1 (NIH)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-08

CONDITIONS: Kyphosis
Keywords: Kyphosis; Yoga; Aging; Physical performance; Quality of Life
MeSH Terms: conditions — Kyphosis | interventions — Yoga; Artifacts; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Yoga, one hour class, 3 times per week, for 24 weeks
  Interventions: Behavioral: Yoga, one hour class, 3 times per week, for 24 weeks
- 2 (Placebo Comparator): Luncheon Seminar Series, once per month, for 24 weeks
  Interventions: Behavioral: Luncheon Seminar Series, once per month, for 24 weeks

INTERVENTIONS:
Behavioral: Yoga, one hour class, 3 times per week, for 24 weeks — Yoga, one hour class, 3 times per week, for 24 weeks
  Arms: 1
Behavioral: Luncheon Seminar Series, once per month, for 24 weeks — Luncheon Seminar Series, once per month, for 24 weeks
  Arms: 2

SUMMARY:
This study seeks to determine whether a specially designed Hatha Yoga program can reduce hyperkyphosis in men and women who are at least 60 years of age and who have excessive thoracic kyphosis.

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or greater
* willingness to accept randomization
* adult-onset hyperkyphosis (noticed after age 50)
* measured Debrunner kyphometer angle >40 degrees

Exclusion Criteria:

active angina; uncontrolled hypertension (SBP greater than 160 or DBP greater than 90); high resting pulse or respiratory rate (HR >90 or RR>24 after 5 minutes seated); current unstable asthma or exacerbated chronic obstructive pulmonary disease; cervical spine instability; unstable knee or shoulder joints; hemiparesis or paraparesis; use of assistive walking device or wheelchair; unable to hear or see adequately for participation in Yoga classes; unable to comprehend and follow directions (in English); unable to attend in-person classes; likely to move within the year after screening; has not had check-up by health care provider within 12 months (if not taking any prescription medications) or in the past 6 months (if any regular medicines taken) and is not willing to do so prior to enrollment; cannot pass physical safety tests. Physical safety was assessed as the ability to stably execute each of the following movements without human assistance: transition from standing to recumbent on the floor and get up from the floor to standing; lift both arms to shoulder level without losing balance; stand with feet side-by-side for 30 seconds; and stand with feet hip-width apart for 60 seconds.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The primary outcomes were change in the following: Debrunner kyphometer-assessed kyphosis angle, standing height, timed chair stands, functional reach and walking speed. | Baseline to 6 months

SECONDARY OUTCOMES:
Secondary outcomes were change in: kyphosis index, flexicurve kyphosis angle, Rancho Bernardo Blocks, pulmonary function and several domains of health-related quality of life (HRQOL). | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gail A Greendale, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Division of Geriatrics, Los Angeles, California, United States